CLINICAL TRIAL: NCT00062010
Title: Interferon Alpha (NSC# 377523) Plus 13-Cis-Retinoic Acid Modulation Of BCL-2 Plus Paclitaxel For Recurrent Small Cell Lung Cancer
Brief Title: Interferon Alfa, Isotretinoin, and Paclitaxel in Treating Patients With Recurrent Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000304430; E6501 (Other: ECOG)
Record Dates: First submitted 2003-06-05; First posted 2003-06-06 (Estimated); Results first posted 2013-01-04 (Estimated); Last update posted 2023-07-07 (Actual); Status verified 2023-06

CONDITIONS: Lung Cancer
Keywords: recurrent small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Small Cell Lung Carcinoma | interventions — Interferon-alpha; Introns; Isotretinoin; Paclitaxel; Taxes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IFN-alpha, 13-CRA, paclitaxel (Experimental): Interferon alpha: 6 million U/m2 on days 1 and 2 of each week for 6 weeks of an 8-week cycle 13-cis-retinoic acid: 1 mg/kg on days 1 and 2 of each week for 6 weeks of an 8-week cycle Paclitaxel: 75 mg/m2 on day 2 of each week for 6 weeks of an 8-week cycle
  Interventions: Biological: interferon alpha; Drug: 13-cis-retinoic acid; Drug: paclitaxel

INTERVENTIONS:
Biological: interferon alpha — Interferon alpha given subcutaneously, 6 million units per square meter of body surface area on days 1 and 2 of each week for 6 weeks, followed by 2 weeks of rest. Given until disease progression or unacceptable toxicity.
  Other Names: Interferon Alpha-2b; Intron-A; IFN-alpha 2b; NSC# 377523
Drug: 13-cis-retinoic acid — 13-cis-retinoic acid given at 1 mg/kg of body weight by mouth on days 1 and 2 of each week for 6 weeks, followed by 2 weeks of rest. Given until disease progression or unacceptable toxicity.
  Other Names: Isotretinoin; RO-43,780; Accutane; Cistane
Drug: paclitaxel — paclitaxel administered intravenously with premedication at 75 mg/m2 of body surface area on day 2 of each week for 6 weeks, followed by 2 weeks of rest. Given until disease progression or unacceptable toxicity.
  Other Names: Taxol; NSC #125973

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as paclitaxel, work in different ways to stop tumor cells from dividing so they stop growing or die. Some tumors become resistant to chemotherapy drugs. Giving interferon alfa and isotretinoin together with paclitaxel may reduce resistance to the drug and allow the tumor cells to be killed.

PURPOSE: This phase II trial is studying how well giving interferon alfa and isotretinoin together with paclitaxel works in treating patients with recurrent small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the frequency and duration of response in patients with recurrent small cell lung cancer treated with interferon alfa, isotretinoin, and paclitaxel.
* Determine the toxic effects of this regimen in these patients.
* Determine the duration of survival in patients treated with this regimen.
* Correlate the levels of bcl-2 in peripheral blood monocytes with response and survival in patients treated with this regimen.

OUTLINE: This is a multicenter study.

Patients receive interferon alfa subcutaneously and oral isotretinoin on days 1 and 2 and paclitaxel IV over 1 hour on day 2 of weeks 1-6. Courses repeat every 8 weeks in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 2 years and then every 6 months for 1 year.

PROJECTED ACCRUAL: A total of 37-83 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria

* Histologically or cytologically confirmed recurrent small cell lung cancer (SCLC) with clinically confirmed measurable disease
* Age 18 and over
* ECOG Performance status 0-3
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Bilirubin no greater than 1.5 mg/dL
* AST no greater than 2 times upper limit of normal (ULN)
* Creatinine no greater than 1.5 mg/dL
* Triglycerides no greater than 1.5 times ULN
* Patients must have had prior chemotherapy treatment for SCLC, and toxicities must have resolved to less than or equal to grade 1
* Women of childbearing potential and sexually active males are strongly encouraged to use an accepted and effective method of contraception.

Exclusion Criteria

* History of another neoplasm other than SCLC except for non-metastatic, non-melanoma skin cancers, carcinoma in situ of the cervix, or cancer cured by surgery or small field radiotherapy at least 5 years before registration
* Pregnant or nursing, with a negative pregnancy test within 2 weeks prior to registration
* Severe depression requiring medication
* Use of the following drugs within 4 weeks prior to registration: carbamazepine, ethanol, tetracycline, doxycycline, minocycline, topical acne products containing Retin-A, vitamin A, cisplatin, ketoconazole, phenytoin or other antiepileptic drugs
* Use of GM-CSF or G-CSF within 4 weeks prior to registration
* Prior paclitaxel or interferon therapy
* Radiation therapy within 60 days prior to registration
* Chemotherapy within 60 days prior to registration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2004-05-26 (Actual); Primary Completion 2011-05 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Aisner, MD, Study Chair — Rutgers Cancer Institute of New Jersey
Locations (73):
- United States (73):
  - Veterans Affairs Medical Center - Atlanta (Decatur), Decatur, Georgia
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - Hinsdale Hematology Oncology Associates, Hinsdale, Illinois
  - Joliet Oncology-Hematology Associates, Limited - West, Joliet, Illinois
  - Swedish-American Regional Cancer Center, Rockford, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Elkhart General Hospital, Elkhart, Indiana
  - Howard Community Hospital, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Saint Joseph Regional Medical Center, South Bend, Indiana
  - Mercy Capitol Hospital, Des Moines, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - McCreery Cancer Center at Ottumwa Regional, Ottumwa, Iowa
  - Borgess Medical Center, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Lakeland Regional Cancer Care Center - St. Joseph, Saint Joseph, Michigan
  - Duluth Clinic Cancer Center - Duluth, Duluth, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - Miller - Dwan Medical Center, Duluth, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Meeker County Memorial Hospital, Litchfield, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - HealthEast Cancer Care at St. Joseph's Hospital, Saint Paul, Minnesota
  - St. Francis Cancer Center at St. Francis Medical Center, Shakopee, Minnesota
  - HealthEast Cancer Care at Woodwinds Health Campus, Woodbury, Minnesota
  - Cancer Resource Center - Lincoln, Lincoln, Nebraska
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - CCOP - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Hunterdon Regional Cancer Center at Hunterdon Medical Center, Flemington, New Jersey
  - CCOP - Northern New Jersey, Hackensack, New Jersey
  - Our Lady of Mercy Medical Center Comprehensive Cancer Center, The Bronx, New York
  - Akron City Hospital, Akron, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Case Comprehensive Cancer Center, Cleveland, Ohio
  - MetroHealth Cancer Care Center at MetroHealth Medical Center, Cleveland, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Grant Medical Center Cancer Care, Columbus, Ohio
  - Mount Carmel Health - West Hospital, Columbus, Ohio
  - Doctors Hospital at Ohio Health, Columbus, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - St. Rita's Medical Center, Lima, Ohio
  - Strecker Cancer Center at Marietta Memorial Hospital, Marietta, Ohio
  - Licking Memorial Cancer Care Program at Licking Memorial Hospital, Newark, Ohio
  - Mercy Medical Center, Springfield, Ohio
  - Community Hospital of Springfield and Clark County, Springfield, Ohio
  - Mount Carmel St. Ann's Cancer Center, Westerville, Ohio
  - Genesis - Good Samaritan Hospital, Zanesville, Ohio
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Cancer Center of Paoli Memorial Hospital, Paoli, Pennsylvania
  - CCOP - MainLine Health, Wynnewood, Pennsylvania
  - Lankenau Cancer Center at Lankenau Hospital, Wynnewood, Pennsylvania
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Medical X-Ray Center, PC, Sioux Falls, South Dakota
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - West Virginia University - Robert C. Byrd Health Sciences Center - Charleston Division, Charleston, West Virginia
  - Mary Babb Randolph Cancer Center at West Virginia University Hospitals, Morgantown, West Virginia
  - Gundersen Lutheran Cancer Center at Gundersen Lutheran Medical Center, La Crosse, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from ECOG member institutions between February 24, 2004 and August 22, 2007. The first patient was accrued on May 26, 2004.
Groups:
- IFN Alpha, 13-Cis-RA, Paclitaxel: Interferon alpha and 13-cis-retinoic acid given on days 1 and 2 and paclitaxel given on day 2 for six weeks of an eight-week cycle until disease progression or unacceptable toxicity
Period: Overall Study
Arm/Group | IFN Alpha, 13-Cis-RA, Paclitaxel
Started | 37
Eligible and Treated | 34
Completed | 34
Not Completed | 3
Not completed — Ineligible | 3

BASELINE CHARACTERISTICS:
Groups:
- IFN 13CRA Paclitaxel: Interferon alpha and 13-cis-retinoic acid given on days 1 and 2 and paclitaxel given on day 2 for six weeks of an eight-week cycle until disease progression or unacceptable toxicity
Arm/Group | IFN 13CRA Paclitaxel
Number analyzed (Participants) | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 26
  >=65 years | 8
Age, Continuous [Median (Full Range); unit: years] | 60 [39 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 22
Region of Enrollment [Number; unit: participants]
  United States | 34

OUTCOME MEASURES:

1. Primary Outcome: Response by RECIST Criteria (v 1.0)
Description: Number of eligible, treated participants in each response category by RECIST criteria
Time Frame: Assessed every 6 weeks
Population: Eligible, treated patients
Measure: Number; unit: participants
Arm/Group | IFN 13CRA Paclitaxel
Number analyzed (Participants) | 34
participants
  Partial Response | 3
  Stable Disease | 5
  Progressive Disease | 11
  Unevaluable | 15
Statistical Analysis 1: Comparison: IFN 13CRA Paclitaxel; The study was designed to have adequate (90%) power to distinguish a true response rate of 50% from a null rate of 35% assuming total accrual of 76 patients in two stages. The design mandated that at least 13 objective responses be observed among 34 patients in the first stage in order to continue to the second stage. These were not observed, so the study stopped after the first stage. 90% exact binomial confidence intervals are provided for the response rate; Test type: Superiority or Other; Overall Response Percentage = 8.8, 90% CI 2-sided [2.4 to 21.3]

2. Secondary Outcome: Survival
Description: Time from registration to death.
Time Frame: Assessed every 3 months for 1 year then every 6 months
Population: Eligible, treated patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | IFN 13CRA Paclitaxel
Number analyzed (Participants) | 34
months | 6.2 [4.7 to 9.8]

3. Secondary Outcome: Progression-free Survival
Description: Time from registration to documented disease progression (RECIST criteria) or death.
Time Frame: Assessed every 6 weeks
Population: Eligible, treated patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | IFN 13CRA Paclitaxel
Number analyzed (Participants) | 34
months | 2.0 [1.8 to 3.9]

ADVERSE EVENTS:
Time Frame: Assessed weekly during treatment
Groups:
- IFN Alpha, 13-CRA, Paclitaxel: Interferon alpha and 13-cis-retinoic acid given on days 1 and 2 and paclitaxel given on day 2 for six weeks of an eight-week cycle until disease progression or unacceptable toxicity
Arm/Group | IFN Alpha, 13-CRA, Paclitaxel
Serious Adverse Events (participants affected / at risk) | 21/34
Other Adverse Events (participants affected / at risk) | 33/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IFN Alpha, 13-CRA, Paclitaxel (N=34)
Leukopenia (Blood and lymphatic system disorders) | 11
Neutropenia (Blood and lymphatic system disorders) | 8
Transfusion-Red Blood Cells (Blood and lymphatic system disorders) | 2
Hypotension (Vascular disorders) | 1
Fatigue (General disorders) | 7
Dehydration (Metabolism and nutrition disorders) | 2
Dysphagia (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Alkaline Phosphatase Increased (Investigations) | 1
AST Increased (Investigations) | 1
ALT Increased (Investigations) | 1
Febrile Neutropenia (Investigations) | 1
Infection with Grade 3 or 4 Neutropenia (Infections and infestations) | 1
Infection without Neutropenia (Infections and infestations) | 1
Amylase Increased (Investigations) | 1
Hypertriglyceridemia (Metabolism and nutrition disorders) | 4
Hypokalemia (Metabolism and nutrition disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 1
Lipase Increased (Investigations) | 1
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 2
"Neuropathy, Motor" (Nervous system disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | IFN Alpha, 13-CRA, Paclitaxel (N=34)
Lymphopenia (Blood and lymphatic system disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 13
Edema (General disorders) | 4
Fever (General disorders) | 7
Rigors/Chills (General disorders) | 14
Sweating (Skin and subcutaneous tissue disorders) | 2
Weight Loss (Investigations) | 6
Constitutional (General disorders) | 2
Prothrombin Time Increased (Investigations) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 11
Dry Skin (Skin and subcutaneous tissue disorders) | 5
Pruritus (Skin and subcutaneous tissue disorders) | 3
Rash/Desquamation (Skin and subcutaneous tissue disorders) | 3
Anorexia (Metabolism and nutrition disorders) | 12
Constipation (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 2
Mouth Dryness (Gastrointestinal disorders) | 5
Nausea (Gastrointestinal disorders) | 8
Stomatitis (Gastrointestinal disorders) | 4
Taste Disturbance (Nervous system disorders) | 6
Diarrhea (Gastrointestinal disorders) | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Bilirubin Increased (Investigations) | 5
Hyperglycemia (Metabolism and nutrition disorders) | 2
Hypomagnesemia (Metabolism and nutrition disorders) | 2
Confusion (Psychiatric disorders) | 2
Dizziness/Lightheadedness (Nervous system disorders) | 4
Insomnia (Psychiatric disorders) | 3
Depression (Psychiatric disorders) | 4
Neuropathy, Sensory (Nervous system disorders) | 11
Pain, Abdominal (Gastrointestinal disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 11
Pain, Bone (Musculoskeletal and connective tissue disorders) | 2
Headache (Nervous system disorders) | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 5
Pain, Other (General disorders) | 2
Creatinine Increased (Investigations) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No